CLINICAL TRIAL: NCT04539574
Title: Validation of a Multi-Parametric Ultra-High Field MRI Protocol for Central Nervous System Malignancy
Brief Title: An Investigational Scan (7T MRI) for the Imaging of Central Nervous System Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1032; NCI-2020-06374 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1032 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Central Nervous System Neoplasm; Glioma; Metastatic Malignant Neoplasm in the Central Nervous System; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (7T MRI) (Experimental): Patients undergo 7T MRI over 60 minutes.
  Interventions: Procedure: 7 Tesla Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: 7 Tesla Magnetic Resonance Imaging — Undergo 7T MRI
  Other Names: 7 Tesla MRI; 7T MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial investigates how well 7T MRI scan works in imaging central nervous system tumors. Diagnostic procedures, such as 7T MRI, may help find and diagnose central nervous system tumors and help measure a patient's response to earlier treatment. The goal of this trial is to learn if a new MRI system can provide better quality images than a standard MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the contrast-to-noise ratio (CNR) for several imaging modalities in brain malignancy as compared with normal brain parenchyma separately by type of malignancy and treatment status.

SECONDARY OBJECTIVE:

I. To assess the conspicuity of each imaging modality to differentiate radiation necrosis from progressive disease.

EXPLORATORY OBJECTIVES:

I. To assess patient experience in the 7 Tesla (7T) magnetic resonance imaging (MRI) system compared to their most recent MRI examination.

II. To assess the typical significance values seen for areas of maximal brain activity associated with each functional MRI (fMRI) test.

III. To assess the geometric distortion of a radiation planning sequence on a ultra-high field (UHF) system.

OUTLINE:

Patients undergo 7T MRI over 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients must meet one set of inclusion criteria:

  * Newly identified and untreated central nervous system glioma or metastasis of at least 5 mm or greater in size

    * Suspected central nervous system neoplasms will require agreement from a study neuroradiologist and a study neurosurgeon or a radiation oncology that a lesion exists that is most likely either a glioma or a metastasis
    * Patients with suspected brain metastasis must also have a history of solid organ malignancy
  * History of central nervous system glioma or metastasis treated with surgery, radiation, chemotherapy, or immunotherapy with new or increasing signal on MR imaging that is suspicious for progressive disease (treatment failure)

    * Suspected recurrent neoplasms will require agreement from a study neuroradiologist and a study neurosurgeon, radiation oncologist, or neuro-oncologist that lesion behavior is suspicious for recurrent disease

Exclusion Criteria:

* Contraindication to MR imaging
* Absolute or relative contra-indication to 3T MRI due to metallic foreign bodies and devices and/or other conditions that are not MR safe, which include implants with unknown behavior in 3T MRI as well as:

  * Electronically, magnetically, and mechanically activated implants
  * Ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers
  * Metallic splinters in the eye
  * Ferromagnetic hemostatic clips in the central nervous system (CNS) or body
  * Cochlear implants
  * Other pacemakers, e.g., for the carotid sinus
  * Insulin pumps and nerve stimulators
  * Non-MR safe lead wires
  * Prosthetic heart valves (if dehiscence is suspected)
  * Non-ferromagnetic stapedial implants
* Pregnancy
* Claustrophobia that does not readily respond to oral medication
* Known allergy to gadolinium-based contrast agents
* Renal failure as defined by a glomerular filtration rate (GFR) less than 30 or the use of hemodialysis
* Pregnant
* Interval treatment with radiation or surgery between the diagnostic MRI lesion identification and planned study MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Wintermark, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 13 years old and above with newly identified and untreated primary brain tumor or metastasis of at least 5 mm or greater in size. Up to twenty (20) healthy volunteers will be studied for the purposes of MRI sequence optimization
Groups:
- Group 1: Healthy Volunteers
- Group 2: Patients (13 years old and above)
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 8 | 30
Completed | 8 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 8 | 30 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 24 | 32
  >=65 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 18 | 23
  Male | 3 | 12 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 27 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 8 | 30 | 38

OUTCOME MEASURES:

1. Primary Outcome: Contrast-to-noise Ratio (CNR)
Description: Contrast-to-noise ratio (CNR) refers to the difference in signal intensity between the tumor and surrounding tissue. Higher CNR values indicate better image quality.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: contrast-to-noise ratio
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 30
contrast-to-noise ratio | 60.6 (26.6) | 58.4 (28.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/30
Other Adverse Events (participants affected / at risk) | 0/8 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04539574/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04539574/ICF_001.pdf